CLINICAL TRIAL: NCT06521775
Title: Pilot Study Evaluating PSMA PET For Metastatic Adenoid Cystic Carcinoma
Brief Title: An Investigational Scan (Ga-68 PSMA-11 PET/CT) for the Detection of Therapy Response in Patients With Metastatic Adenoid Cystic Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-003306; NCI-2024-05893 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-003306 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-07-19; First posted 2024-07-26 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Adenoid Cystic Carcinoma
MeSH Terms: conditions — Carcinoma, Adenoid Cystic | interventions — gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (Ga-68 PSMA-11, PET/CT) (Experimental): Patients receive Ga-68 PSMA-11 IV and then undergo PET/CT 50-70 minutes after injection at baseline and approximately 12-20 weeks during investigational therapy.
  Interventions: Procedure: Computed Tomography; Other: Electronic Health Record Review; Drug: Ga-68 PSMA-11; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Other: Electronic Health Record Review — Ancillary studies
Drug: Ga-68 PSMA-11 — Given IV
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-DKFZ-PSMA-11; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA; 68Ga-PSMA-11; 68Ga-PSMA-HBED-CC; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; AAA 517; AAA-517; AAA517; Ga PSMA; Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled PSMA-11; Gallium Ga 68 PSMA-11; Gallium Ga 68-labeled PSMA-11; GALLIUM GA-68 GOZETOTIDE; Gallium-68 PSMA; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; GaPSMA; PSMA-HBED-CC GA-68; Gallium Ga 68 Gozetotide
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase II trial tests whether gallium-68 (Ga-68) prostate specific membrane antigen (PSMA)-11 positron emission tomography (PET)/computed tomography (CT) imaging is useful for detecting therapy response in patients with adenoid cystic carcinoma (salivary gland cancer) that has spread from where it first started (primary site) to other places in the body (metastatic). The PET scan detects and takes pictures of where the radioactive imaging agent (68Ga PSMA-11) has gone in the body and the CT scan uses x-rays to create images of the bones and internal organs within the body. Combining a PET scan with a CT scan can help make the images easier to interpret. This study may help researchers learn whether GA-68 PSMA-11 PET/CT is useful for detecting treatment response and guiding treatment decisions in patients with metastatic adenoid cystic carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the feasibility of serial Ga-68 PSMA PET/CT for response assessment in metastatic adenoid cystic carcinoma.

II. Assess the correlation of PSMA PET/CT response assessment with serum extracellular vesical (EV) PSMA levels for patients undergoing treatment for metastatic adenoid cystic carcinoma.

OUTLINE:

Patients receive Ga-68 PSMA-11 intravenously (IV) and then undergo PET/CT 50-70 minutes after injection at baseline and approximately 12-20 weeks during investigational therapy.

After completion of study intervention, patients are followed up at 1 day.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Diagnosis of metastatic adenoid cystic carcinoma
* Enrolled in protocol MC200708
* Ability to tolerate a Ga68 PSMA PET/CT imaging study
* Willingness to return for a second PSMA PET/CT scan in approximately 12-20 weeks from the baseline PET/CT
* Ability to give appropriate consent or have an appropriate representative available to do so

Exclusion Criteria:

* Unable to undergo PET/CT scan
* Not a participant in MC200708
* < 18 years of age
* Persons who are pregnant or nursing
* Persons unable to consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Treatment response assessment (Feasibility) | Up to 20 weeks
  Data from the prostate specific membrane antigen (PSMA) positron emission tomography (PET)/computerized tomography (CT) exams will be categorized into treatment response categories for each participant using the Response Evaluation Criteria in PSMA PET/CT (RECIP) 1.0 criteria. Tumor volume with PSMA expression on PET/CT will be quantified using MIM Software Version 7.2.7.
Response assessment category and percent change in tumor volume | Up to 20 weeks
  Will be correlated to percent change in serial PSMA extracellular vesical (EV) from serum measurements from participant data obtained in the MC200708 trial protocol. For continuous measurements (like percent change), scatter plots and simple linear regression will be conducted. Associations of these continuous variables will be done via the Spearman's rank correlation coefficient. For assessment of changes, will use Wilcoxon Signed-Rank test. For any associations of categorical variables, will use the Fisher's Exact test.
Incidence of adverse events | Up to 20 weeks
  Will be assessed by the number of adverse event incidents reported. Safety will be categorized using the the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Percentage change of mean standardized uptake value (SUV) of index lesions | Up to 20 weeks
  Will be correlated with percentage change in PSMA EVs.
Percentage change of PSMA-avid tumor volume | Up to 20 weeks
  Will be assessed on PET correlated with percentage change in PSMA EVs.

CONTACTS AND LOCATIONS:
Overall Officials: Brian J. Burkett, MD, MPH, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials